CLINICAL TRIAL: NCT00919165
Title: Assessment of Cognitive Function in Patients Undergoing Carotid Artery Stent Placement: Cognitive Function in Carotid Stenting
Brief Title: Assessment of Cognitive Function in Patients Undergoing Carotid Artery Stent Placement
Status: Completed | Type: Observational
Sponsor: Corewell Health West (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 2007-286
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Cognitive Function in Carotid Stenting
Keywords: carotid stenting; cognitive function; pre and post stent; severe carotid artery stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- control and study group: severe carotid artery stenosis in asymptomatic patients defined as greater than 80% stenosis angiographically or greater than 400 cm/sec peak systolic velocity on carotid doppler evaluation

SUMMARY:
To determine the effect of carotid artery stenting, on cognitive function, in patients with high grade carotid artery stenosis

DETAILED DESCRIPTION:
Single Center, Case Controlled design using pre and post stent cognitive function testin. Patients will serve as self controls to observe the effect, if any, of carotid stent placement on cognitive function in asymptomatic patients with high grade carotid artery stenosis

ELIGIBILITY:
Inclusion Criteria:

* 40-80 years of age
* Right hand dominate
* Asymptomatic:defined as: no symptoms of TIA/stroke in the previous 6 months
* Baseline doppler study with a peak systolic velocity of 400cm/sec
* Patient is deemed candidate for carotid artery stenting
* TIMI flow of 1,2 or 3
* 80% or greater stenosis of distal common or internal carotid artery, as determined angiographically, as defined in ACAS
* Subjects are able to give informed consent
* Subjects are willing/able to complete follow-up visits

Exclusion Criteria:

* History of major stroke: within the past 6 months
* History of Alzheimers disease or Dementia
* Unable or willing to complete the baseline and 20 days neuro-cognitive testing planned major surgery within the next 2 months
* Planned intervention opposite carotid artery within 2 months
* Ineligibility for carotid stent procedure due to anatomy, thrombus, or inability to complete anti-platelet therapy
* Any individual identified with cognitive impairment which would affect their performance during cognitive testing.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe carotid artery stenosis
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2007-12; Primary Completion 2017-03 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
to determine the effect of carotid artery stenting, on cognitive function after carotid artery stenting in patients with severe carotid artery stenosis | 45 days

SECONDARY OUTCOMES:
to evaluate the clinical benefit of carotid artery stenting on cognitive function, pre and post carotid artery stenting | 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Steven Pastyrnak, PhD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States